CLINICAL TRIAL: NCT03011918
Title: Eat Well, Fall Less
Brief Title: Malnutrition's Role in Fall Risk
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary M. Julius, RD,CDE, Research Dietitian Nutritionist, Louis Stokes VA Medical Center
Other Study IDs: 13009-H06
Record Dates: First submitted 2015-08-31; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Falling Injury; Nutrition Disorder
MeSH Terms: conditions — Nutrition Disorders | interventions — Vitamin D; C-Reactive Protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observational Single Event Faller: one documented fall as an in-patient. It is hypothesized that the nutrition factors present prior to the first fall may be related to fall frequency. Data on exposure to nutrition supplementation will be collected for future analysis. Subpopulation alalysis of individuals with dementia will also be conducted
  Interventions: Other: Data Collection prior to first fall for all fallers; Other: Hgb value; Other: Vitamin D; Other: C-Reactive Protein
- Observational Multiple event faller: multiple falls documented during in-patient stay It is hypothesized that frequent fallers will demonstrate statistically greater weight decline, Hgb decline, Vitamin D deficiency and Higher C-Reactive Protein values prior to the first fall. Data on exposure to nutrition supplementation will be collected for future analysis.. Subpopulation analysis of individuals with dementia will also be conducted.
  Interventions: Other: Data Collection prior to first fall for all fallers; Other: Hgb value; Other: Vitamin D; Other: C-Reactive Protein

INTERVENTIONS:
Other: Data Collection prior to first fall for all fallers — Weight history. Descriptive analysis of weight history in single event fallers compared to multiple event fallers. Information on use of any nutrition supplementation exposure will also be collected
  Other Names: percent weight loss
Other: Hgb value — Hgb decline. Descriptive analysis of single event fallers compared to multiple event fallers will be analyzed. Use of nutrition supplement exposure will be collected
Other: Vitamin D — Descriptive analysis of vitamin D status of single event fallers compared to multiple event fallers will be analyzed. Use of nutrition supplement exposure will be collected..
Other: C-Reactive Protein — Descriptive analysis of C-RP value status of single event fallers as compared to multiple event fallers will be analyzed. Use of nutrition supplement exposure data will be collected.

SUMMARY:
Falls and falls related injuries are considered one of the most adverse events that a patient can experience. Several assessment instruments to assess and mitigate risks for falls have been developed. However, these instruments have not addressed nutritional risk factors.

Weight loss and low hemoglobin levels are key components of Malnutrition. Malnutrition in the hospital setting is a significant concern and may play a role as a fall risk factor.

The World Health Organization (WHO) maintains a global anemia database. WHO has identified iron deficiency anemia, based on hemoglobin value alone as the most common, wide-spread nutritional deficiency worldwide. Anemia is present in 30% of the worlds population including industrialized nations.

The consensus statement of the Academy of Nutrition and Dietetics / American Society of Parenteral and Enteral Nutrition simply defines adult under-nutrition as a continuum of inadequate intake along with a multitude of other factors. Weight loss occurs at multiple points along this continuum.

this multiphase retrospective descriptive analysis hypothesizes that degree of weight loss and degree of Hgb decline may be fall risk factors.

DETAILED DESCRIPTION:
Eat Well, Fall Less is a multiphase retrospective descriptive analysis of single event fallers and repeat fallers. Data source: Documented falls occurring between October 1, 2010 and October 31, 2012.

Chart Review data on weight loss and decline in Hemoglobin levels were collected 12 months, 6 months and 3months and 1 month prior to the first fall along as the most recent value prior to the event. Additional data on vitamin D levels and C-reactive Protein values will be collected at the 12 month, 6month, and 1 month prior to the first fall

Statistical Analysis using SAS version 9.1. a two tailed t-test was performed to evaluate differences in HGB characteristics between single and frequent fallers. One way ANOVA evaluated changes in Hgb, c-Reactive Protein, vitamin D values and weight over time are being collected.

Two constellations of fallers emerged. Those with and those without dementia. The two groups appeared to have different nutrition risk factors. All statistical analysis was done using JMP Pro (version 10.0.0, SAS Institute, Inc, Cary, NC). Statistical significance was set at p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Veteran experienced a fall during a hospitalization between October 1, 2010 and October 31, 2012
* Veteran must have at least one documented weight a minimum of 24 months prior to admission

Exclusion Criteria:

* Adults who suffer from neurological disease or stroke
* Adults with documented orthopedic fracture in the past 12 months
* Documented amputation of a lower limb in the past 24 months
* Blindness
* History of volume overload, renal, cardiovascular or other in nature
* current alcoholic
* It is felt that a co-morbidity exists which makes the individuals weight history inaccurate, such as a recent prosthetic device alteration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized veterans having experiencced a fall between october 31, 2010 nad October 31, 2012
Sampling Method: Non-Probability Sample
Enrollment: 485 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Eat Well, Fall Less | 4 year
  Multiphase descriptive analysis

CONTACTS AND LOCATIONS:
Locations (1):
- LSCVAMed Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be made available to future dietitians and Geriatric researchers obtaining an IRB approved protocol for ad hoc analysis.